CLINICAL TRIAL: NCT04173468
Title: Comparison of Mobilization With Movement and Mulligan Knee Taping Technique on Patellofemoral Pain Syndrome.
Brief Title: Mobilization With Movement Versus Mulligan Knee Taping Technique on Patellofemoral Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Mubara Rehman
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Patellofemoral Syndrome
Keywords: Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Movement

STUDY DESIGN:
Intervention Model Description: There will be two groups of participant. One group will receive MWM along with conventional therapy and the second group group will receive Mulligan knee taping along with conventional therapy.
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWM Group (Active Comparator): This group will receive Mobilization with Movement (MWM) i.e. straight leg raised with traction,Tibial Gliding
  Interventions: Other: Moblization with Movement
- Mulligan Taping Group (Active Comparator): This group will receive Mulligan knee taping
  Interventions: Other: Mulligan knee taping

INTERVENTIONS:
Other: Moblization with Movement — patients with group 1 will receive two techniques pertaining to MWM intervention (straight leg raised with traction and tibial Gliding) Repeat it 10 times,3 sets and 1 mint interval. .For Tibial Gliding we will asks the patient to perform 10 repetitive active knee extensions. Practice will be performed by doing 10 reps for 3 sets with 1 min interval. After this home exercises will b guided stretching of hamstrings 8 to 10 reps 20 sec hold, strengthening of Quadriceps and VMO with 10 reps and 3 sets
  Arms: MWM Group
Other: Mulligan knee taping — patient with group 2 will receive Mulligan taping technique. Tape will be applied for two days then we will change it. After this home based exercise will be guided which is stretching of hamstrings 8 to 10 reps 20 sec hold , strengthening of Quadriceps and VMO with 10 reps and 3 sets.
  Arms: Mulligan Taping Group

SUMMARY:
This study intends to determine the effects of MWM verses Mulligan knee taping on patellofemoral pain syndrome.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial, will be conducted at Pakistan railway general hospital Rawalpindi. Both MWM and Mulligan knee taping Techniques are used in patients with patellofemoral pain syndrome. Sample size of 34 individuals was calculated through Open Epi tool version 3 with 95 % confidence interval (CI), and power 80%. 34 individuals were screened out on the basis of inclusion and exclusion criteria. Individuals of this selected population were randomly allocated as 17 individuals in MWM (straight leg raise with traction and tibial gliding) group and 17 individuals Mulligan knee taping group by sealed envelope method. And after this Both groups will receive conventional therapy.

Assesment will be done at baseline, 2nd week and after 6 weeks Data will be analyzed on SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:• Anterior knee Pain durations lasting longer than two months,

* Pain scoring three or more according to Numeric pain Rating scale (NPRS) during at least two activities
* Age between 20 and 45 years
* Both Genders

Exclusion Criteria:

* • Past history of total knee artthroplasty

  * Intra articular steroid injection
  * Rheumatoid Arthritis
  * Use of Assistive devices e.g. canes, walkers and braces
  * Knee injury

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Time up and Go test | Baseline
  Patients were asked to perform test at usual walking speed .initial testing standardized verbal instruction given to the participant regarding procedure. For performing TUG participants were instructed to walk three meter and then walk back to sit down .Note time on stopwatch .The average of tests trail was measured as the mean of TUG.
Time up and Go test | Post 2nd week
  Patients were asked to perform test at usual walking speed .initial testing standardized verbal instruction given to the participant regarding procedure. For performing TUG participants were instructed to walk three meter and then walk back to sit down .Note time on stopwatch .The average of tests trail was measured as the mean of TUG.
Time up and Go test | Post 6 week
  Patients were asked to perform test at usual walking speed .initial testing standardized verbal instruction given to the participant regarding procedure. For performing TUG participants were instructed to walk three meter and then walk back to sit down .Note time on stopwatch .The average of tests trail was measured as the mean of TUG.
Active knee extension test | Baseline
  Active knee extension test (AKE), is used to assess hamstring length. It was performed while the participant was in supine lying and involved leg was in 90 degree hip flexion. Then participant was asked to extend the knee. For hamstring tightness cut off score AKE angle is 160°. Therefore normal individuals with angle < 160° were considered as individuals with hamstring tightness. Its reliability is 0.94.
Active knee extension test:(2nd week) | Post 2nd Week
  Active knee extension test (AKE), is used to assess hamstring length. It was performed while the participant was in supine lying and involved leg was in 90 degree hip flexion. Then participant was asked to extend the knee. For hamstring tightness cut off score AKE angle is 160°. Therefore normal individuals with angle < 160° were considered as individuals with hamstring tightness. Its reliability is 0.94.
Active knee extension test:(6 week) | Post 6th Week
  Active knee extension test (AKE), is used to assess hamstring length. It was performed while the participant was in supine lying and involved leg was in 90 degree hip flexion. Then participant was asked to extend the knee. For hamstring tightness cut off score AKE angle is 160°. Therefore normal individuals with angle < 160° were considered as individuals with hamstring tightness. Its reliability is 0.94.
Sit and reach Test | Baseline
  Sit and reach test (SRT) is most commonly employed test to measure hamstring flexibility. This tool is used to measure range of hamstring muscle at knee joint.Each participant was instructed to sits on a couch in long sitting position. participants were seated with elongated legs, with hip flexed to 90 degrees and knees were fully extended and the ankles were in relaxed plantar flexion. A measuring ruler/tape was placed,between the feet with 38 cm score was marked tangent to the sole of the feet. Subjects were asked to reach forward with hands one above the other and palms of the hands facing down, while attempting to touch fingertips to toes or as far beyond on measuring tape while keeping the knees straight.
Sit and reach Test | Post 2nd week
  Sit and reach test (SRT) is most commonly employed test to measure hamstring flexibility. This tool is used to measure range of hamstring muscle at knee joint.Each participant was instructed to sits on a couch in long sitting position. participants were seated with elongated legs, with hip flexed to 90 degrees and knees were fully extended and the ankles were in relaxed plantar flexion. A measuring ruler/tape was placed,between the feet with 38 cm score was marked tangent to the sole of the feet. Subjects were asked to reach forward with hands one above the other and palms of the hands facing down, while attempting to touch fingertips to toes or as far beyond on measuring tape while keeping the knees straight.
Sit and reach Test( 6 week) | Post 6th Week
  Sit and reach test (SRT) is most commonly employed test to measure hamstring flexibility. This tool is used to measure range of hamstring muscle at knee joint.Each participant was instructed to sits on a couch in long sitting position. participants were seated with elongated legs, with hip flexed to 90 degrees and knees were fully extended and the ankles were in relaxed plantar flexion. A measuring ruler/tape was placed,between the feet with 38 cm score was marked tangent to the sole of the feet. Subjects were asked to reach forward with hands one above the other and palms of the hands facing down, while attempting to touch fingertips to toes or as far beyond on measuring tape while keeping the knees straight.

SECONDARY OUTCOMES:
NPRS Numeric Pain Rating Scale | Baseline
  (NPRS)is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric Pain Rating Scale (NPRS) [ 2nd week] | Post 2nd week
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric Pain Rating Scale (NPRS) [ 6th week ] | Post 6th Week
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Kujala pain Rating score:(Baseline) | Baseline
  The Kujala pain rating scale is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. For example, a 'Limp' score would be scored as follows: none (5), slight/periodic (3), constant (0). Total scores range from 0 to 100.
Kujala pain Rating scale : (2nd week) | Post 2nd week
  The Kujala pain Rating scale [ is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. For example, a 'Limp' score would be scored as follows: none (5), slight/periodic (3), constant (0). Total scores range from 0 to 100
Kuala pain Rating Scale: (6th week) | Post 6th week
  The kujala pain rating scale is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. For example, a 'Limp' score would be scored as follows: none (5), slight/periodic (3), constant (0). Total scores range from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demirci S, Kinikli GI, Callaghan MJ, Tunay VB. Comparison of short-term effects of mobilization with movement and Kinesiotaping on pain, function and balance in patellofemoral pain. Acta Orthop Traumatol Turc. 2017 Dec;51(6):442-447. doi: 10.1016/j.aott.2017.09.005. Epub 2017 Oct 17. PMID 29054803
- [Background] Hickey A, Hopper D, Hall T, Wild CY. The Effect of the Mulligan Knee Taping Technique on Patellofemoral Pain and Lower Limb Biomechanics. Am J Sports Med. 2016 May;44(5):1179-85. doi: 10.1177/0363546516629418. Epub 2016 Feb 22. PMID 26903215
- [Background] Callaghan MJ, Selfe J. Patellar taping for patellofemoral pain syndrome in adults. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD006717. doi: 10.1002/14651858.CD006717.pub2. PMID 22513943